CLINICAL TRIAL: NCT03415932
Title: Health Group Intervention Among Refugees in Sweden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Pia Yngman-Uhlin, Principal investigator, Region Östergötland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20117278-31
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Migration Stress

STUDY DESIGN:
Intervention Model Description: baseline and follow up in one population
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health education (Experimental): Assessment of healt care Contacts Before and after intervention
  Interventions: Behavioral: health education

INTERVENTIONS:
Behavioral: health education — Health information by a multimodal team

SUMMARY:
This prospective intervention study evaluates whether health education and basic body awareness training reduces health care consumption and improves movement quality among refugees in Sweden.

DETAILED DESCRIPTION:
Migration is well known to be stressful and to have a negative impact on Health. Multidisciplinary health-promoting group interventions have significantly improved self-rated health. Further, symptom improvement was shown after implementation of physical activity in form of basic body awareness training. In this study a multimodal team consisted of a physiotherapist, nurse, psychologist, dietician, and physician held sessions of three hours weekly for a period of nine weeks. The sessions started with basic body awareness training, followed by theme discussions on symptoms and health strategies. A total of 54 participants completed the intervention. Health care consumption and movement quality were measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria: Refugees seeking primary care consultation or rehabilitation unit aged 18-65 years were candidates for inclusion. Based on the health care provider's assessment, patients whose health symptoms could be connected to or increased by the migration process were eligible for inclusion -

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Health care consumption | three months before and after intervention
  number of Health care contacts

IPD SHARING:
Plan to Share IPD: No